CLINICAL TRIAL: NCT02944526
Title: The Effect of 3 Ropivacaine Suprascapular Nerve Blocks in Subacute Adhesive Capsulitis: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinique Saint-Jean, Bruxelles (Other)
Collaborators: University Hospital St Luc, Brussels (Other)
Responsible Party: Principal Investigator, Marc Schiltz, MD, Dr Marc Schiltz MD, Head of Department Physical Medicine and Rehabilitation, Clinique Saint-Jean, Bruxelles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-10/02
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder; Nerve Block
Keywords: suprascapular nerve
MeSH Terms: conditions — Bursitis | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine Suprascapular Nerve Block (Experimental): Suprascapular nerve block realized in sterile conditions under live ultrasound guidance: injection of 5ml of Ropivacaine monohydrochloride 2mg/ml.
  3 successive blocks are realized at 1 week interval.
  Interventions: Drug: Ropivacaine Monohydrochloride
- Placebo Suprascapular Nerve Block (Placebo Comparator): Suprascapular nerve block realized in sterile conditions under live ultrasound guidance: injection of 5ml of physiological /isotonic saline.
  3 successive blocks are realized at 1 week interval.
  Interventions: Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: Ropivacaine Monohydrochloride — Suprascapular nerve block under ultrasound control: injection of 5ml Ropivacaine HCL 2mg /ml
  Arms: Ropivacaine Suprascapular Nerve Block
Drug: Placebo - Concentrate — Placebo suprascapular nerve block under ultrasound control: injection of 5ml physiological / isotonic saline
  Arms: Placebo Suprascapular Nerve Block

SUMMARY:
Patients presenting with subacute, less than 6 months of evolution, adhesive capsulitis are randomly attributed to the control or study group. Both groups receive a series of 3 suprascapular nerve blocks under ultrasound guidance with either 5ml saline or 5ml ropivacaine 2mg/ml ( ref) at 1 week interval. Testing consists of glenohumeral range of motion (ROM) (anterior elevation, lateral elevation, external and internal rotation) measured by goniometer, Constant score and visual analog scale (VAS) pain score. Evaluations are done immediately before and one hour after every suprascapular block and at 4 weeks after the third suprascapular block.

All suprascapular nerve blocks are performed by one physician and the evaluations are done by a occupational therapist or MD experienced in glenohumeral function evaluations. All practitioners are blinded to the assigned group.

All patients continue their pre-study treatment of physiotherapy and per os pain medication. Patients keep a record of analgesics and NSAID use during the trial. Drop-out rate is measured.

DETAILED DESCRIPTION:
Introduction: Adhesive capsulitis is a painful and debilitating condition affecting adult shoulders. Although relatively rare the condition is more common in diabetic patients and effective pain diminishing treatments without the use of corticosteroids are needed.

Methods and Material: Patients presenting with subacute, less than 6 months of evolution, adhesive capsulitis are randomly attributed to the control or study group. Both groups receive a series of 3 successive suprascapular nerve blocks under live ultrasound guidance with either 5ml saline or 5ml ropivacaine 2mg/ml conducted at 1 week interval. Testing consists of glenohumeral ROM (anterior elevation, lateral elevation, external and internal rotation) measured by goniometer, Constant score, VAS pain score. Evaluations are done immediately before and one hour after every "suprascapular block" and at 4 weeks after the third suprascapular block.

All suprascapular blocks are performed by one physician and the evaluations by either a occupational therapist or MD experienced in glenohumeral function evaluations. All practitioners are blinded to the assigned group.

All patients continue their physiotherapy, consisting of electrotherapy, range of motion, stretching and strengthening exercises and their per os medication. Patients keep record of analgesics and NSAID use during the trial. Drop-out rate is measured during the entire study protocol.

ELIGIBILITY:
Inclusion Criteria:

* subacute adhesive capsulitis: pain evolving for less than 6 months before enrollment

Exclusion Criteria:

* other conditions involving the shoulder ( rheumatoid or septic arthritis, Hill-Sachs lesions,osteoarthritis of the shoulder, or malignancies in the shoulder region);
* neurologic deficits affecting shoulder function in normal daily activities (such as history of stroke, multiple sclerosis, parkinson disease...)
* shoulder pain caused by cervical radiculopathy
* a history of drug allergy to ropivacaïne
* pregnancy or lactation
* cognitive impairment with inability to fill out a protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
change in constant shoulder score | at 0, 1, 2, and 6 weeks
  the total constant score ranges from 0 to 100 points, with higher scores indicative of better function. The score is divided into four sections: pain, activity of daily living, ROM and strength
change of pain intensity score | at 0,1,2 and 6 weeks
  pain intensity measured by visual analog scale (VAS)

SECONDARY OUTCOMES:
change in gleno-humeral joint range of motion (ROM) | at 0,1,2, and 6 weeks
  Shoulder flexion, abduction, external rotation and internal rotation measured with goniometer with the patient in standing position

CONTACTS AND LOCATIONS:
Overall Officials: SCHILTZ Marc, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Marc Schiltz, MD, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No